CLINICAL TRIAL: NCT05772637
Title: Clinical and Urodynamic Assessment of Bladder Sensation in Multiple Sclerosis
Acronym: CUBS-MS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP230079
Record Dates: First submitted 2023-02-22; First posted 2023-03-16 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-02

CONDITIONS: Overactive Bladder
Keywords: overactive bladder; multiple sclerosis; bladder sensations
MeSH Terms: conditions — Urinary Bladder, Overactive; Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MS Patient with Bladder disorders (Experimental)
  Interventions: Procedure: Repeated cystometries with bladder sensations assessment

INTERVENTIONS:
Procedure: Repeated cystometries with bladder sensations assessment — A second cystometry will be performed to assess bladder sensations reliability. A third cystometry with cognitive task (STROOP test) at the same time will be performed to assess the impact of distractive attentional task on bladder sensations

SUMMARY:
The aim of the study is to assess the association between bladder sensations progression during bladder filling and severity of Overactive bladder (OAB) in patients with multiple sclerosis.

DETAILED DESCRIPTION:
Lower urinary tract symptoms (LUTS) are frequent in central nervous system disorders especially in patients with multiple sclerosis (PwMS). Prevalence of LUTS is important (32 to 96.8%) and increases with multiple sclerosis (MS) duration and the severity of the neurological deficiencies and disabilities. Overactive bladder (OAB) with urgency, frequency, urgency urinary incontinence, is the most common symptom, reported by 37-99% of the PwMS. Voiding difficulties are less common, from 6 to 49%, and usually appear later with the course of the disease.

Urodynamics is a useful test recommended to understand the mechanism of bladder dysfunction, and look for risk factors of upper tract damage.

Detrusor overactivity is the most reported mechanism of overactive bladder, and describes the occurrence of uninhibited contractions of the detrusor during bladder filling. But abnormal bladder sensations, with increased or decreased sensations, have also been described. The prevalence of these abnormalities is not well described, however, in the absence of detrusor overactivity, abnormal afferent information (i.e., abnormal bladder sensations) is the plausible mechanism involved in urinary disorders.

The assessment of bladder sensations is still a poorly explored field. Bladder diary can be used for the collection of the intensity of need to void with a Likert scale or numerical scale.

During cystometry, it is recommended to collect different bladder sensations: first sensation of filling, first desire to void, strong desire to void, urgent desire to void. However, it has been described that bladder sensations progress in 8 to 9 different levels of intensity in healthy subjects.

The aim of the study is to assess the association between bladder sensations progression during bladder filling and severity of OAB in patients with multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* MS according to the 2017 Mac Donald diagnostic criteria
* Bladder disorders supposedly related to MS
* Indication to perform urodynamics
* No current medication for bladder disorders
* Able to understand and right in French
* Affiliated to the "Securite sociale" or "Couverture Medicale Universelle (CMU)", or equivalent organism.

Exclusion criteria:

* Legal protection
* Pregnancy or breastfeeding mother
* MS relapse during the past month
* Other associated neurological disease
* Genuine stress incontinence related to postpartum
* Treatment with antimuscarinics, alpha blockers, beta3 adrenergic, or tibial nerve stimulation in the past 15 days, or with botulinic toxin injection in the past 6 months
* Previous lower urinary tract surgery
* Inability to use the analogic device due to motor, sensory or ataxic disabilities

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2025-02-14 (Estimated); Study Completion 2025-02-14 (Estimated)

PRIMARY OUTCOMES:
bladder sensation ( area under the sensation-capacity curve (AUC)) | Day 1
  The areas under the sensation-capacity curve (AUC) will be calculated for individual participants using the trapezoidal rule for specific capacity ranges.

SECONDARY OUTCOMES:
bladder sensitivity | Day 1
  Bladder sensitivity assessed by the number of steps in the evolution of the need to urinate reported by the patient (number of times the cursor of the analogical scale is moved), during the filling.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital TENON, Paris, Choisir Une Région, France

IPD SHARING:
Plan to Share IPD: Undecided